CLINICAL TRIAL: NCT01076621
Title: A 12 Month Non-interventional (Observational), International, Multi-centre, Prospective Study to Evaluate the Bleeding Pattern of Ultra-low Dose Continuous Combined Hormone Replacement Therapy Containing 0.5 mg Estradiol and 0.1 mg Norethisterone Acetate (Eviana®)
Brief Title: Observational Study to Investigate the Occurrence of Bleeding in Postmenopausal Women Treated With Estradiol/NETA for 12 Months
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: ALD-3795; U1111-1112-8626 (Other: WHO)
Record Dates: First submitted 2010-02-25; First posted 2010-02-26 (Estimated); Last update posted 2014-10-27 (Estimated); Status verified 2014-10

CONDITIONS: Menopause; Postmenopausal Bleeding
MeSH Terms: interventions — Estradiol; Norethindrone Acetate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- A
  Interventions: Drug: 0.5 mg estradiol / 0.1 mg norethisterone acetate (NETA)

INTERVENTIONS:
Drug: 0.5 mg estradiol / 0.1 mg norethisterone acetate (NETA) — Data collection of the use of 0.5 mg estradiol and 0.1 mg norethisterone acetate (NETA) in women in connection to a daily clinical practice.

SUMMARY:
This study is conducted in Europe. The primary aim of this observational study is to investigate the occurrence of bleeding in women taking 0.5 mg estradiol and 0.1 mg norethisterone acetate (NETA) for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent, permitting the data to be processed within the scope of the study, is obtained from the patient before any study-related activities
* Postmenopausal amenorrhoeic women
* Treatment with previously combined HRT discontinued at least 3 months prior to start of 0.5 mg estradiol and 0.1 mg norethisterone acetate treatment

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The postmenopausal women (who are ammenorrheic) are to be offered participation in the study at the discretion of the treating physician following the decision to prescribe 0.5 mg estradiol and 0.1 mg norethisterone acetate for the treatment of their menopausal symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 176 (Actual)
Dates: Start 2010-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Bleeding profile during the 52 weeks of treatment with 0.5 mg estradiol and 0.1 mg norethisterone acetate evaluated by bleeding, and bleeding or spotting rates | At every lunar month (28 days)

SECONDARY OUTCOMES:
Change in bleeding profile | During the 52 weeks of treatment
Change in mean number of hot flushes per week | During the 52 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (2):
- Rud, Norway
- Gothenburg, Sweden

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com